CLINICAL TRIAL: NCT01737359
Title: A Phase IIa, Randomized, Double-blind, Active-controlled, 12-week Study of Amdoxovir (Two Doses) Versus Tenofovir DF, in Combination With Zidovudine in HIV-1 Treatment-experienced Subjects With M184I/V Mutation in Addition to 0-2 Confirmed Thymidine Analog Mutations.
Brief Title: A Safety and Efficacy Study of Amdoxovir in HIV-1 Treatment-experienced Subjects.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: RFS Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RFSP-AMDX-2010
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2013-03

CONDITIONS: Human Immunodeficiency Virus Infection
Keywords: amdoxovir; zidovudine; tenofovir DF; HIV; HAART; antiretroviral
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — amdoxovir; BID protein, human; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- amdoxovir 300 mg bid (Experimental): in combination with zidovudine 300 mg bid for 12 weeks; lopinavir/ritonavir (400 mg/100 mg) bid is added on week 3
  Interventions: Drug: amdoxovir 300 mg bid
- amdoxovir 500 mg bid (Experimental): in combination with zidovudine 300 mg bid for 12 weeks; lopinavir/ritonavir (400 mg/100 mg) bid is added on week 3
  Interventions: Drug: amdoxovir 500 mg bid
- tenofovir DF 300 mg qd (Active Comparator): in combination with zidovudine 300 mg bid for 12 weeks; lopinavir/ritonavir (400 mg/100 mg) bid is added on week 3
  Interventions: Drug: tenofovir DF 300 mg qd

INTERVENTIONS:
Drug: amdoxovir 300 mg bid — 2 x 150 mg capsules bid
  Other Names: DAPD; AMDX
  Arms: amdoxovir 300 mg bid
Drug: amdoxovir 500 mg bid — 2 x 250 mg capsules bid
  Other Names: DAPD; AMDX
  Arms: amdoxovir 500 mg bid
Drug: tenofovir DF 300 mg qd — 1 x 300 mg tablet once daily
  Other Names: Viread
  Arms: tenofovir DF 300 mg qd

SUMMARY:
This is a double-blind Phase 2a study to test the safety and efficacy of an investigational HIV drug, amdoxovir (300 mg or 500 mg twice daily) compared with tenofovir DF 300 mg once daily in HIV-1 infected antiretroviral therapy-experienced subjects who are currently failing antiretroviral therapy. There are three treatment groups (N=45). Subjects will be randomized to receive either amdoxovir 300 mg twice daily (n=15) or amdoxovir 500 mg twice daily (n=15) or tenofovir DF 300 mg once daily (n=15); each in combination with zidovudine 300 mg twice daily.

The study will assess initially amdoxovir (300 mg or 500 mg twice daily) or tenofovir DF 300 mg once daily, both in combination zidovudine 300 mg twice daily plus failing third drug, but then with lopinavir/ritonavir (400 mg/100 mg twice daily) after Week 2. Subjects who received amdoxovir (300 mg or 500 mg twice daily) and benefited from the drug may choose to enroll in the 36-week open-label study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years old with HIV-1 RNA ≥ 2,000 copies/mL and currently failing therapy.
* Has M184I/V mutation in addition to 0-2 thymidine analog mutations (TAMs) at screening.
* Agree to be abstinent or use two reliable forms of contraception (for females) and one form for men when participating in sexual activity that could result in pregnancy.

Exclusion Criteria:

* Current or recent (last 30 days of study entry) AIDS defining diseases.
* Genotypic resistance testing at screening indicating K65R, L74V, Q151M mutation.
* Prior exposure to lopinavir/ritonavir or amdoxovir.
* Impaired hepatic function (ALT > 5 x ULN).
* Women who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
HIV-1 viral load | change from baseline to Week 2
Safety and Tolerability- Incidence of adverse events and laboratory abnormalities | number and frequency from baseline through Week 12

SECONDARY OUTCOMES:
HIV-1 viral load | change from baseline to Weeks 4, 8 and 12
Changes in Immunologic Function (CD4 cell counts) | changes from baseline to Weeks 4, 8 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Luz Pascual, MD MPH, Study Director — RFS Pharma
Locations (2):
- Argentina (2):
  - Research Site, Buenos Aires, Buenos Aires
  - Research Site, Rosario, Santa Fe Province